CLINICAL TRIAL: NCT00769431
Title: FOCUS GROUP EVALUATION OF PROSTATE CANCER SYMPTOM MANAGEMENT EDUCATION MATERIALS
Brief Title: Evaluating Symptom Management Educational Materials for Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, David Latini, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CDR0000600594; BCM-H-21622
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Focus group (No Intervention)
  Interventions: Other: educational intervention; Other: study of socioeconomic and demographic variables

INTERVENTIONS:
Other: educational intervention
Other: study of socioeconomic and demographic variables

SUMMARY:
RATIONALE: Collecting feedback from patients with prostate cancer may help doctors develop better symptom management educational materials for patients.

PURPOSE: This clinical trial is evaluating symptom management educational materials for patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To collect formative evaluation data about a new educational intervention using focus groups of patients with prostate cancer.
* To use the focus group data in the master's research paper of a Baylor College of Medicine physician-assistant student who is documenting the process of organizing and conducting the focus groups, enumerating areas where the new materials are deemed problematic, and identifying themes in the comments made by the focus group participants.

OUTLINE: Study participants are assigned to 1 of 3 focus groups according to educational level and ethnicity (i.e., lower educational-level African-American men primarily from the Michael E. DeBakey Veterans Affairs Medical Center (MEDVAMC); lower educational-level Caucasian men from MEDVAMC, Baylor College of Medicine (BCM), or the community; or higher educational-level Caucasian men primarily from BCM or the community).

Participants review written patient educational-intervention materials on prostate cancer and provide feedback to the investigator on the content and acceptability of these materials during a 1½-2-hour focus group discussion. Feedback data are used to revise the intervention materials so that they are appropriate to the target population.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven prostate cancer

  * Localized disease that has been previously treated
* Selected for participation from 1 of the following:

  * Convenience sample of men from the Baylor College of Medicine (BCM) Urology clinics at Scurlock Tower (including the Urology clinic at MEDVAMC) and local prostate cancer-support groups
  * Prostate cancer survivors who participated in the US TOO Father's Day Walk/Run or the Gay Pride Celebration

PATIENT CHARACTERISTICS:

* Able to speak and read in English
* Willing to review the written patient educational materials and discuss them in a group setting

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Acceptability of the written patient educational materials, in terms of text size, white space, font, and graphics | Single timepoint
Formative evaluation of the new educational materials, in terms of the comments made by the focus group participants | Single timepoint
Validation that the goals of the educational-intervention instruction are being achieved | Single timepoint
Improvement of the educational-intervention instruction by identification and remediation of problems | Single timepoint

CONTACTS AND LOCATIONS:
Overall Officials: David M. Latini, PhD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas